CLINICAL TRIAL: NCT00888212
Title: Minimally Invasive Techniques Or Surgery In the Diagnosis of Sarcoidosis (MITOSIS-Trial)
Brief Title: Minimally Invasive Techniques Or Surgery In the Diagnosis of Sarcoidosis
Acronym: MITOSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Kurt Tournoy, MD, PhD, University Hospital Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008/069
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchoscopy (Experimental): Bronchoscopy, only if no diagnosis is obtained, patients go for EUS-FNA or EBUS-TBNA, only if no diagnosis is obtained, patients go for surgical biopsy
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopy, only if no diagnosis is obtained, patients go for EUS-FNA or EBUS-TBNA, only if no diagnosis is obtained, patients go for surgical biopsy

SUMMARY:
The purpose of this study is to evaluate the yield of endoscopic guided fine needle aspirations (by means of transoesophageal endoscopic ultrasound : EUS-FNA or transbronchial endoscopic ultrasound : EBUS-TBNA) in patients with a clinical suspicion for sarcoidosis stage I-II; but in whom the preceding bronchoscopy did not result in a qualifying diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 y
* Suspicion of thoracic sarcoidosis and need for tissue confirmation
* Recent (<6 weeks) RX and CT-thorax (HRCT not compulsory)
* Fit for bronchoscopy (with or without EBB, TBB, TBNA), esophagoscopy and surgery
* Written informed consent

Exclusion Criteria:

* Patients with obvious other organ involvement allowing "simple and safe" biopsy
* Lofgren syndrome
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The diagnostic yield of state-of-the art bronchoscopy (including TBB, EBB and TBNA) | At the end of study
The role of endosonography (EUS-FNA or EBUS-TBNA) in demonstrating non-caseating granulomas after a non-qualifying bronchoscopy | At the end of study

SECONDARY OUTCOMES:
Prevalence of sarcoidosis and alternate diagnosis | At the end of study
Stage distribution | At the end of study
Complication rate of each type of procedure | At the end of study
Cost to obtain a qualifying diagnosis with this strategy in this population | At the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Kurt G. Tournoy, Md, PhD, Principal Investigator — University Hospital, Ghent
Locations (15):
- Belgium (14):
  - OLV Ziekenhuis Aalst, Aalst
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - ZNA Antwerpen, Antwerp
  - AZ St. Jan Hospitaal Brugge, Bruges
  - Cliniques Universitaires St. Luc, Brussels
  - Höpital Erasme Brussel, Brussels
  - University Hospital Brussels, Brussels
  - CHU Charleroi, Charleroi
  - University Hospital Ghent, Ghent
  - Virga Jesse Hospitaal, Hasselt
  - UZ Gasthuisberg Leuven, Leuven
  - Heilig Hartziekenhuis Menen, Menen
  - Hôpital Saint Elisabeth Namur, Namur
  - AZ Oudenaarde, Oudenaarde
- Ampha Ziekenhuis Breda, Breda, Netherlands

REFERENCES:
- [Derived] Tournoy KG, Bolly A, Aerts JG, Pierard P, De Pauw R, Leduc D, Leloup A, Pieters T, Slabbynck H, Janssens A, Carron K, Schrevens L, Pat K, De Keukeleire T, Dooms C. The value of endoscopic ultrasound after bronchoscopy to diagnose thoracic sarcoidosis. Eur Respir J. 2010 Jun;35(6):1329-35. doi: 10.1183/09031936.00111509. Epub 2009 Nov 6. PMID 19897553
- See also: Website of the University Hospital Ghent — http://www.uzgent.be